CLINICAL TRIAL: NCT04142385
Title: Incidence of Human Immunodeficiency Virus (HIV) Among Indian Men Who Have Sex With Men (MSM)
Brief Title: Incidence of HIV Infection in Screening Indian Men Who Have Sex With Men
Status: Withdrawn | Type: Observational
Why Stopped: Closed due to lack of funding.
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Tata Memorial Hospital (Other Government); Udaan Trust (Unknown); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-093; NCI-2016-01358 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-093; AMC-093 (Other: AIDS Malignancy Consortium); AMC-093 (Other: CTEP); R21CA167652 (NIH); UM1CA121947 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-10-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Independent Medical Evaluation; Restraint, Physical; Proctoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (health information collection): Participants receive a questionnaire, undergo a targeted physical and anal clinical exam, undergo blood collection and urethral swab for STIs, and a penile skin cell and anal swab for cytology and HPV DNA at months 0, 6, and 12. Participants also undergo HRA and penile clinical exam at month 12.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Medical Examination; Procedure: Physical Examination; Procedure: Proctoscopy with Biopsy; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo blood, urethral swab, penile skin cell, and anal swab collection
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Medical Examination — Undergo anal and penile clinical exam
  Other Names: Exam; Examination; Medical Assessment; Medical Exam; Medical Inspection
Procedure: Physical Examination — Undergo targeted physical exam
  Other Names: Assessment; Physical; Physical Assessment; Physical Exam
Procedure: Proctoscopy with Biopsy — Undergo HRA
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the incidence of human immunodeficiency virus (HIV) infection in screening Indian men who have sex with men (MSM). Gathering health information over time from Indian MSM may help doctors determine how many Indian MSM develop new cases of HIV infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the one-year incidence of HIV among high-risk MSM in India.

SECONDARY OBJECTIVES:

I. To test the feasibility and acceptability of recruiting a sample of 150 high-risk HIV-uninfected MSM using respondent-driven sampling (RDS) and following them every six months for one year.

II. To produce preliminary descriptive data on the prevalence and incidence of human papillomavirus (HPV) infection and HPV-associated disease and sexually transmitted infections (STIs) other than HPV in HIV-seronegative MSM in India.

III. To produce preliminary descriptive data on sexual risk behaviors with men and women, as well as data on other potential confounders.

OUTLINE:

Participants receive a questionnaire, undergo a targeted physical and anal clinical exam, undergo blood collection and urethral swab for STIs, and a penile skin cell and anal swab for cytology and HPV deoxyribonucleic acid (DNA) at months 0, 6, and 12. Participants also undergo high-resolution anoscopy (HRA) and penile clinical exam at month 12.

ELIGIBILITY:
Inclusion Criteria:

* HIV seronegative, as documented by any licensed HIV test according to National Acquired Immunodeficiency Syndrome (AIDS) Control Organization (NACO) guidelines
* Participants report any sex with a man in the past 6 months
* Participants must speak Hindi, Marathi, or English
* Participant should not have any plans to move out of the area in the next 12 months and commit to attending two additional visits one at 6 months and one at 12 months

Exclusion Criteria:

* Active drug or alcohol use or dependence, or other impairment that, in the opinion of the site investigator, would interfere with adherence to study requirements

  * Participants with impairments that, in the opinion of the site Investigator, are temporary, will be asked to return another day for enrollment
* Inability to provide informed consent
* History of a sex change operation that would preclude collection of penile or scrotal specimens

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-seronegative MSM in Mumbai, India
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2027-04-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of human immunodeficiency virus (HIV) | Up to 12 months
  The total number of participants with incident HIV divided by the total follow-up will be used to calculate the incidence per 100 person years. HIV status is determined by HIV rapid test and a confirmatory Western blot test.

SECONDARY OUTCOMES:
Successful respondent-driven sampling (RDS) | 3 months
  Defined as half of the study sample enrolled and at least 50% of the responses to the questions of RDS acceptability are answered "Not at all embarrassed or burdened by RDS".
Successful respondent-driven sampling (RDS) | 12 months
  Defined as more than 80% of participants recruited through RDS.
Prevalence of penile human papillomavirus (HPV) infection, assessed by polymerase chain reaction (PCR) | Up to 12 months
  Summarized using proportions and exact 95% binomial confidence interval (CI). Will be estimated for specific types and for all combined.
Prevalence of human papillomavirus (HPV)-associated lesions of the penis | Up to 12 months
  Summarized using proportions and exact 95% binomial CI. Will be estimated for specific types and for all combined.
Prevalence of human papillomavirus (HPV)-associated lesions of the anus | Up to 12 months
  Summarized using proportions and exact 95% binomial CI. Will be estimated for specific types and for all combined.
Prevalence of anal human papillomavirus (HPV) infection, assessed by polymerase chain reaction (PCR) | Up to 12 months
  Summarized using proportions and exact 95% binomial confidence interval (CI). Will be estimated for specific types and for all combined.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, Principal Investigator — AIDS Malignancy Consortium
Locations (3):
- UCSF Medical Center-Parnassus, San Francisco, California, United States
- India (2):
  - Tata Memorial Hospital, Mumbai
  - Udaan Trust, Mumbai

IPD SHARING:
Plan to Share IPD: Undecided